CLINICAL TRIAL: NCT05844696
Title: Electrical Neuromodulation for Focal Epilepsy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202207164DINA
Record Dates: First submitted 2023-04-11; First posted 2023-05-06 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham stimulation (Sham Comparator)
  Interventions: Device: Soterix MXN-5 HD-tES Model 5005A. Medtronic Percept DBS platform.
- continuous tDCS (Experimental)
  Interventions: Device: Soterix MXN-5 HD-tES Model 5005A. Medtronic Percept DBS platform.
- slow-oscillatory tDCS (Experimental)
  Interventions: Device: Soterix MXN-5 HD-tES Model 5005A. Medtronic Percept DBS platform.

INTERVENTIONS:
Device: Soterix MXN-5 HD-tES Model 5005A. Medtronic Percept DBS platform. — 〔Part 1〕Using Soterix MXN-5 HD-tES Model 5005A. Three treatment groups: sham control, continuous tDCS, slow-oscillatory tDCS.
  〔Part 2〕Using Medtronic Percept DBS platform. Single group:Neuromodulation.

SUMMARY:
The purpose of this research is to use electrical neuromodulation on patients with focal epilepsy. The main objective is to assess safety and observe potential therapeutic effects.

ELIGIBILITY:
Inclusion Criteria:

Part 1

* Age ≥ 20 years old.
* Focal epilepsy patients having received EEG and brain imaging studies and on standard medication.

Part 2

* Age ≥ 20 years old.
* Focal epilepsy patients having received EEG and brain imaging studies and on standard medication for at least 1 year.
* Having received part I intervention.

Exclusion Criteria:

Part 1

* Patients with secondary and progressive macrostructural abnormalities in the brain, such as brain tumors or infectious lesions. This does not include abnormalities directly related to epilepsy, such as mesial temporal sclerosis or focal dysplasia.
* Patients who are unable to undergo brain electrical stimulation, including those with metal in the brain or implanted stimulators/implants.
* Patients with allergies to the sponge material used for stimulation.
* Patients with wounds or infections at the site of sponge application.
* Patients with intellectual disabilities, manic episodes (with a score of greater than 12 on the Young Mania Rating Scale), major physiological illnesses (such as stroke, brain tumors, or heart attacks), or pregnant or breastfeeding women.
* Patients judged by the physician to be unsuitable for the clinical trial due to unstable vital signs or serious internal or external medical conditions.

Part 2

* Patients with secondary and progressive macrostructural abnormalities in the brain, such as brain tumors or infectious lesions. This does not include abnormalities directly related to epilepsy, such as mesial temporal sclerosis or focal dysplasia.
* Patients who could be considered for single focus resection based on the neurologist/neurosurgeon's judgment. However, patients who clearly refuse resection surgery are not subject to this limitation.
* Patients who experience serious adverse events (SAEs) during the part 1 trial.
* Patients who are unable to undergo magnetic resonance imaging (MRI).
* Patients who are planned to receive hyperthermia therapy or transcranial magnetic stimulation.
* Patients judged by the physician to be unsuitable for the clinical trial due to unstable vital signs or serious internal or external medical conditions.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 3 months
  Any noxious, unintended and undesired effect

SECONDARY OUTCOMES:
The seizure frequency per month | 3 months
  Seizure per month

IPD SHARING:
Plan to Share IPD: No